CLINICAL TRIAL: NCT02844608
Title: Quality of Life Assessment in Routine Clinical Oncology Practice at the University Hospital of Besancon
Brief Title: Feasibility of Quality of Life Assessment in Routine Clinical Oncology Practice at the University Hospital of Besancon
Acronym: QOLIBRY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2015/274
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer
Keywords: Health-related quality of life; Oncology clinical practice; Electronic collection
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quality of Life (Other): Administration of Quality of Life questionnaires
  Interventions: Other: Quality of Life Questionnaires

INTERVENTIONS:
Other: Quality of Life Questionnaires — Patients will be asked to complete standardized HRQoL questionnaires: the EORTC QLQ-C30 with its specific module by cancer site (QLQ-BR23, QLQ-CR29, QLQ-LC13) at first visit before starting treatment and then before every medical consultation during four months.

SUMMARY:
Symptoms related to the disease and/or treatment are common in cancer patients and can affect patient health-related quality of life (HRQol). Unfortunately these symptoms can be underestimated and underreported by the physician. Measure of the HRQoL has been significantly developed in clinical trials and has become a key endpoint to assess clinical benefit of new therapeutic strategies and as prognostic factor of overall survival for several cancer as in women breast cancer, glioblastomas, metastatic colorectal cancer, prostate cancer and hepatocellular carcinoma.

Moreover, a recent study conducted in patients receiving routine outpatient chemotherapy for advanced solid tumors showed that clinical benefits were associated with symptom self-reporting during cancer care, including the improvement of the overall survival.

The aim of the QOLIBRY project is to introduce the collection of HRQoL of cancer patients in daily clinical practice in the University Hospital of Besançon. Indeed, the goal is to make the HRQoL data accessible and exploitable in real time to physician, to help medical professionals to optimize their practices by adopting a holistic and personalized approach based on the perception of the patients of their HRQoL and symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of using in routinely clinical practice a systematic assessment of HRQoL in patients treated for a newly diagnosis cancer at the University Hospital of Besançon. It aims to define the logistic resources needed to implement this data collection and to assess its acceptability by clinicians, healthcare team and patients. This involves asking patients to complete HRQoL questionnaires at the time of an outpatient visit and generating a summary of the results made available to the healthcare provider immediately before the consultation.

In this pilot study, three cancer sites were selected: breast cancer in women, colorectal cancer and lung cancer. Patients included will be invited to complete the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 cancer specific questionnaire and the specific module of their cancer site (QLQ-BR23, QLQ-CR29, QLQ-LC13) before each visit with their physician. Results from HRQoL questionnaires will be immediately available to physician through a web-based portal during the visit. As part of the pilot phase, patients will be followed during four months while HRQoL will be pursued.

Questionnaires completion will be administrated by digital tablets and/or computer terminals via the CHES software (Computer-based Health Evaluation System; http:// www.ches.pro/) at the University Hospital of Besançon just before the visit with physician or at home via secured web-portal. This tool provides a didactic and attractive presentation of the HRQOL evaluation allowing physician a better understanding and consideration of HRQoL results. Indeed, results of a routinely assessment of HRQoL will be incorporated into the patient's electronic medical record. Physicians will be alerted if a clinically significant deterioration of at least one HRQoL dimension is observed over time and/or if the HRQoL level is significantly lower than reference/ normative data. In case of deterioration of HRQoL, physician may adapted the treatment or prescribed adapted supportive cares.

This feasibility study aims to assess the acceptability of the HRQoL assessment in routinely practice: to quantify the attrition, to observe the exhaustiveness of the measure, the compliance and the ability of the patient to complete HRQoL questionnaires and finally to evaluate both patient and clinician's satisfaction. The difficulties eventually encountered by the clinical research associate and by physicians will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, ≥ 18 years of age
* No prior diagnosis of cancer
* Patients with newly diagnosed breast, colorectal or lung cancer
* No prior therapy for cancer except surgery
* Patients treated at University Hospital of Besançon
* Patients had given their informed consent to participate.

Exclusion Criteria:

* Patients with tumor recurrence,
* Patients with second cancer
* Patients with psychopathology or serious cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-11-10 (Estimated); Study Completion 2019-03-10 (Estimated)

PRIMARY OUTCOMES:
Rate of HRQOL questionnaire completion | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier régional Universitaire de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Velikova G, Booth L, Smith AB, Brown PM, Lynch P, Brown JM, Selby PJ. Measuring quality of life in routine oncology practice improves communication and patient well-being: a randomized controlled trial. J Clin Oncol. 2004 Feb 15;22(4):714-24. doi: 10.1200/JCO.2004.06.078. PMID 14966096
- [Background] Velikova G, Awad N, Coles-Gale R, Wright EP, Brown JM, Selby PJ. The clinical value of quality of life assessment in oncology practice-a qualitative study of patient and physician views. Psychooncology. 2008 Jul;17(7):690-8. doi: 10.1002/pon.1295. PMID 18033733
- [Background] Holzner B, Giesinger JM, Pinggera J, Zugal S, Schopf F, Oberguggenberger AS, Gamper EM, Zabernigg A, Weber B, Rumpold G. The Computer-based Health Evaluation Software (CHES): a software for electronic patient-reported outcome monitoring. BMC Med Inform Decis Mak. 2012 Nov 9;12:126. doi: 10.1186/1472-6947-12-126. PMID 23140270
- [Background] Fromme EK, Eilers KM, Mori M, Hsieh YC, Beer TM. How accurate is clinician reporting of chemotherapy adverse effects? A comparison with patient-reported symptoms from the Quality-of-Life Questionnaire C30. J Clin Oncol. 2004 Sep 1;22(17):3485-90. doi: 10.1200/JCO.2004.03.025. PMID 15337796
- [Background] Fisch MJ, Lee JW, Weiss M, Wagner LI, Chang VT, Cella D, Manola JB, Minasian LM, McCaskill-Stevens W, Mendoza TR, Cleeland CS. Prospective, observational study of pain and analgesic prescribing in medical oncology outpatients with breast, colorectal, lung, or prostate cancer. J Clin Oncol. 2012 Jun 1;30(16):1980-8. doi: 10.1200/JCO.2011.39.2381. Epub 2012 Apr 16. PMID 22508819
- [Background] Seow H, Sussman J, Martelli-Reid L, Pond G, Bainbridge D. Do high symptom scores trigger clinical actions? An audit after implementing electronic symptom screening. J Oncol Pract. 2012 Nov;8(6):e142-8. doi: 10.1200/JOP.2011.000525. Epub 2012 Aug 21. PMID 23598849
- [Background] Kroenke K, Krebs EE, Wu J, Yu Z, Chumbler NR, Bair MJ. Telecare collaborative management of chronic pain in primary care: a randomized clinical trial. JAMA. 2014 Jul 16;312(3):240-8. doi: 10.1001/jama.2014.7689. PMID 25027139
- [Background] Gilbert JE, Howell D, King S, Sawka C, Hughes E, Angus H, Dudgeon D. Quality improvement in cancer symptom assessment and control: the Provincial Palliative Care Integration Project (PPCIP). J Pain Symptom Manage. 2012 Apr;43(4):663-78. doi: 10.1016/j.jpainsymman.2011.04.028. PMID 22464352
- [Background] Valderas JM, Kotzeva A, Espallargues M, Guyatt G, Ferrans CE, Halyard MY, Revicki DA, Symonds T, Parada A, Alonso J. The impact of measuring patient-reported outcomes in clinical practice: a systematic review of the literature. Qual Life Res. 2008 Mar;17(2):179-93. doi: 10.1007/s11136-007-9295-0. Epub 2008 Jan 4. PMID 18175207
- [Background] Berry DL, Blumenstein BA, Halpenny B, Wolpin S, Fann JR, Austin-Seymour M, Bush N, Karras BT, Lober WB, McCorkle R. Enhancing patient-provider communication with the electronic self-report assessment for cancer: a randomized trial. J Clin Oncol. 2011 Mar 10;29(8):1029-35. doi: 10.1200/JCO.2010.30.3909. Epub 2011 Jan 31. PMID 21282548
- [Background] Diouf M, Chibaudel B, Filleron T, Tournigand C, Hug de Larauze M, Garcia-Larnicol ML, Dumont S, Louvet C, Perez-Staub N, Hadengue A, de Gramont A, Bonnetain F. Could baseline health-related quality of life (QoL) predict overall survival in metastatic colorectal cancer? The results of the GERCOR OPTIMOX 1 study. Health Qual Life Outcomes. 2014 May 13;12:69. doi: 10.1186/1477-7525-12-69. PMID 24886671
- [Background] Mauer M, Stupp R, Taphoorn MJ, Coens C, Osoba D, Marosi C, Wong R, de Witte O, Cairncross JG, Efficace F, Mirimanoff RO, Forsyth P, van den Bent MJ, Weller M, Bottomley A. The prognostic value of health-related quality-of-life data in predicting survival in glioblastoma cancer patients: results from an international randomised phase III EORTC Brain Tumour and Radiation Oncology Groups, and NCIC Clinical Trials Group study. Br J Cancer. 2007 Aug 6;97(3):302-7. doi: 10.1038/sj.bjc.6603876. Epub 2007 Jul 3. PMID 17609661